CLINICAL TRIAL: NCT07087483
Title: Effects of a Nurse-Led Transition to Fatherhood Program on Fathers' Involvement in Infant Care, Gender Perception, and Father-Infant Bonding: A Randomized Controlled Trial
Brief Title: Effects of a Nurse-Led Transition to Fatherhood Program on Fathers' Involvement in Infant Care, Gender Perception, and Father-Infant Bonding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University Hospital (Other)
Responsible Party: Principal Investigator, Sati Koldas Mir, Principal Investigator, Akdeniz University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AU-SBF-SKM-01
Record Dates: First submitted 2025-06-26; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Training Effectiveness; Fatherhood Transition Training for New Fathers
Keywords: fathers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The fathers who receive training (Experimental): We will provide a training to fathers how they can improve and support their fatherhood skills with their newborns.
  Interventions: Behavioral: The fathers who receive training; Behavioral: Fatherhood Skill Training
- The fathers who do not receive any training (No Intervention)

INTERVENTIONS:
Behavioral: The fathers who receive training — We will provide training to fathers on how they can improve and support their fatherhood skills with their newborns, and the control group will only receive the brochure about the basic fatherhood skills.
  Arms: The fathers who receive training
Behavioral: Fatherhood Skill Training — FATHERHOOD TRANSITION TRAINING PROGRAM • Explanation of the goals and objectives of the training
  * Introduction to the training program
  * Newborn's physiological characteristics (weight, height, head circumference, fontanelles, body temperature, sleep, feeding, urination, meconium, genital organs, reflexes, sleeping position, safety, hygiene)
  * Infant feeding and burping the baby
  * Changing baby's clothes, giving a bath, diapering, and general care of the eyes, ears, mouth, umbilical cord, and skin
  * Importance and benefits of breast milk
  * Breastfeeding positions and techniques
  * Methods of expressing, storing, and increasing breast milk
  * Information about vaccinations, hearing and heel-prick screening, developmental hip dysplasia, and jaundice
  * General information on gender roles
  * Importance of father-infant bonding and its short- and long-term outcomes
  Arms: The fathers who receive training

SUMMARY:
Fatherhood transition programs led by nurses can positively influence fathers' involvement in infant care, gender roles, and father-infant bonding. These programs encourage fathers to take a more active role in both the prenatal and postnatal periods, enhancing their knowledge and skills related to infant care. Through these programs, fathers gain more information and practical abilities in caring for their babies.

The trainings provided by nurses cover essential care topics such as infant and maternal nutrition, sleep routines, diapering, burping, hygiene, and safety. This knowledge enables fathers to participate in infant care more effectively and safely.

Traditional gender roles often assume that infant care is primarily the mother's responsibility. However, nurse-led programs emphasize that fathers can and should take an active role in this process. This helps break down stereotypes related to gender roles and strengthens the father's role in childcare.

Active participation in infant care from an early stage contributes to the development of a strong emotional bond between father and baby. Quality time spent together, physical contact, and shared activities reinforce this bond. Research shows that a strong father-infant bond has positive effects on a child's emotional and social development.

In conclusion, nurse-led fatherhood transition programs significantly contribute to reshaping traditional gender roles and strengthening the emotional bond between fathers and their babies by increasing paternal involvement in infant care. Expanding such programs can lead to long-term positive outcomes for both fathers and children.

ELIGIBILITY:
Inclusion Criteria:

* being a newborn father

Exclusion Criteria:

* N/A

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Father-Infant Attachment Scale (FIAS) | 0 - 4 months
  The scale, developed by Condon and colleagues, aims to assess father-infant attachment within the first year postpartum (Condon et al., 2008). The Turkish adaptation was conducted by Güleç and Kavlak (2013) and administered to fathers of infants aged 6-12 months. With the author's approval, it was stated that the scale could be used from the third month postpartum onward. The scale consists of 18 items and has three subdimensions: pleasure in interaction, love and pride, and patience and tolerance. Each item on the scale is rated on a scale from 1 to 5. Except for items 1, 2, 3, 6, 17, 18, and 19, the items are reverse-scored. Scoring for reverse items is performed in the opposite direction. Higher scores indicate stronger attachment (Güleç & Kavlak, 2013). A validity and reliability analysis was conducted to evaluate the appropriateness of the scale. At the sixth month, the total Cronbach's alpha coefficient of the scale was determined as 0.81; for the patience and tolerance subdimen

SECONDARY OUTCOMES:
Gender Perception Scale | 0 - 4 months
  Developed by Altınova and Duyan (2013), the Gender Perception Scale, for which validity and reliability studies have been conducted, was designed particularly for use with adults. It measures individuals' attitudes regarding how they perceive gender roles in various areas. This scale consists of a total of 25 items. Ten of the items are positively worded, and fifteen are negatively worded. The scale uses a five-point Likert format, where individuals indicate their level of agreement with the statements as follows: "strongly agree (5), agree (4), undecided (3), disagree (2), strongly disagree (1)." Negative items are reverse-scored. Items 2, 4, 6, 9, 10, 12, 15, 16, 17, 18, 19, 20, 21, 24, and 25 are negative and are reverse-scored. Accordingly, scores on the scale can range between 25 and 125, with higher scores indicating a more positive perception of gender roles. The Cronbach's alpha coefficient of the scale was found to be 0.872.

OTHER OUTCOMES:
Infant Care Interview Form | 0 - 4 months
  Prepared by the researcher in line with the literature (Maraşlı, 2019; Bal, 2014), this form consists of 17 questions covering practices that fathers can individually perform in relation to infant care. It will be administered as both a pre-test and a post-test. this will be used for showing the change in their skills before and after the training

IPD SHARING:
Plan to Share IPD: Undecided
We will ask the participants if they would like to share any details about their participation. upon agreement, the IPD might be considered to share